CLINICAL TRIAL: NCT04615169
Title: Multi-component Cognitive Intervention for Older Adults With Mixed Cognitive Abilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng Kung University (Other)
Responsible Party: Principal Investigator, Ling-Hui Chang, Associate Professor, National Cheng Kung University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: National Cheng Kung University
Record Dates: First submitted 2020-10-23; First posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-10

CONDITIONS: Cognitive Training; Dementia; Occupational Therapy; Aging; Long Term Care
Keywords: cognitive training; dementia prevention; Dementia; occupational therapy; community based practice; older people; long term care
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: A multi-center one-group pretest, post-test, and 3-month follow up design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- multi-component cognitive intervention using simulated everyday tasks (MCI-SET) (Experimental): the 12-week intervention, 2 hours weekly session of MCI-SET.
  Interventions: Behavioral: Multi-component cognitive intervention with simulated everyday tasks (MCI-SET)

INTERVENTIONS:
Behavioral: Multi-component cognitive intervention with simulated everyday tasks (MCI-SET) — 2 hours per session: consisted primarily of modified everyday cognitive tasks, which were adjusted for individuals and for the group by the group leader to provide an error-reduction learning environment. Each session consisted of: (1) Warm-up: a 15-30 minute dual task of motor-cognitive exercises that increase arousal level and provide cognitive stimulation. For example, at the beginning of the group, the members would sing a song, mimic dance movement of the group leader, and clap hands when specific words occur in the song.
  (2) 30-minutes guided and repetitive practices of contextually-relevant simulated everyday cognitive tasks with one 15 to 20- minute break in between; Cognitive tasks addressed complex attention, visual scanning, auditory attention, visual and motor memory, auditory memory, prospective memory, executive functioning, problem solving, etc.

SUMMARY:
Objective: To assess the feasibility and preliminary effectiveness of an evidence-driven, pragmatic multi-component cognitive intervention with simulated everyday tasks (MCI-SET) with an inclusive group design in community centers Methods: One group, pre-test, post-test, and 3-month follow up research design. The participants who were >=65 and frail, dependence in >= one activity of daily living, or with a confirmed dementia from eight community centers. MCI-SET consisted 12 two-hour weekly group sessions. Feasibility was described with intervention development, fidelity, and acceptability. Outcomes included general daily functioning, general cognition, memory, attention, executive functioning, and processing speed.

DETAILED DESCRIPTION:
According to the World Alzheimer Report 2018, 50 million people are living with dementia and the number is expected to triple to 152 million by 2050. Most people at high risk of dementia or with dementia reside in the community. Effective community-based programs can help to maintain functional levels and mitigate or prevent excessive functional decline. There are increasing empirical evidence to support structured and regular cognitive activities as part of brain health lifestyle .

Cognitive intervention is an increasing popular approach that aim to maintain or improve the cognitive functioning of the older adults with or without cognitive impairments. Appropriate cognitive intervention has the potential to change their brain neuro-mechanism. Recent evidence suggests that repeated practices of a carefully designed cognitive exercises with a high degree of similarity with real-life activities of daily living (ADL) (e.g., remembering the instructions for taking prescription medicine, identifying the medicine precautions, etc.) can improve both cognitive skills and cognitive functional performance.

Because of the complexity of cognitive issues people with cognitive impairments encounter, scholars have advocated for a multi-component cognitive intervention that includes more than one approach to make the best use of the individual approaches. The investigators conducted a quasi-experimental study that combined motor-cognitive dual-task exercises with high cognitive demands, cognitive training, and cognitive rehabilitation. The results showed that the intervention can improve cognitive skills and cognitive functional performance for people with mild cognitive impairments.

However, the need to strengthen the research design and to standardize treatment protocols led most cognitive intervention research to target a group of participants with similar cognitive skills, such as those with normal cognition, those with mild cognitive impairments, or those with dementia, etc. This homogeneity in participants is in sharp contrast to what is observed in communities, where most likely the group is inclusive of persons with different levels of cognitive skills. The efficacy of cognitive intervention with an inclusive group design was rarely examined.

Scholars have called for more effort to speed up the process of bridging evidence-based intervention to the everyday settings people live in. Cognitive intervention is in a situation of "leaky pipeline," that is, no systematic examination of how the evidence can be translated, tested in real-world settings (practice), and/or implemented across communities in the continuum of research evidence to widespread implementation. The increasing use of feasibility research design is mostly used as a precursor of randomized clinical trial, examining whether a study protocol requires adjustment, what the barriers and potential strategies are. With the abundance of research that supports the efficacy of cognitive intervention, to the best of the investigators' knowledge, there are no study that investigated the transportability of evidence-based cognitive intervention into the community.

This study discusses the feasibility, implementation, and preliminary effectiveness of an evidence-driven, multi-component cognitive intervention using simulated everyday tasks (MCI-SET) for cognitively-vulnerable older adults in community organizations in two cities in southern Taiwan.

ELIGIBILITY:
Inclusion Criteria:

equal to or more than 65 years old, and frailty status according to the Study of Osteoporotic Fractures (SOF) criteria of frailty, or dependence with at least one daily activities.

Exclusion Criteria:

People with non-cognitive issues, such as severe visual, hearing, or physical impairments, that interfered with completion of evaluations.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 140 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Kihon Checklist-Taiwan (KCL) | up to one month before the start of intervention
  KCL is a self-reported questionnaire, consisted of 25 items (yes/no) divided into 7 sub-categories: general independence, physical strength, nutrition, oral function, level of social activities outside of home, cognitive function, and risk of depression. It takes about 15 minutes to complete. Each item is rated as pass (0) or fail (1). A higher total score indicates worse functioning. KCL has been used as a reliable indicator of daily functioning and progression of disability in Japan National Long-term Care. Taiwan Ministry of Health and Welfare adopted KCL-Taiwan version as an indicator of daily functioning for the use of national-wide disability prevention and delay community-based programs.
Kihon Checklist-Taiwan (KCL) | up to one month after the end of intervention
  KCL is a self-reported questionnaire, consisted of 25 items (yes/no) divided into 7 sub-categories: general independence, physical strength, nutrition, oral function, level of social activities outside of home, cognitive function, and risk of depression. It takes about 15 minutes to complete. Each item is rated as pass (0) or fail (1). A higher total score indicates worse functioning. KCL has been used as a reliable indicator of daily functioning and progression of disability in Japan National Long-term Care. Taiwan Ministry of Health and Welfare adopted KCL-Taiwan version as an indicator of daily functioning for the use of national-wide disability prevention and delay community-based programs.
Kihon Checklist-Taiwan (KCL) | up to 4 months after the end of intervention
  KCL is a self-reported questionnaire, consisted of 25 items (yes/no) divided into 7 sub-categories: general independence, physical strength, nutrition, oral function, level of social activities outside of home, cognitive function, and risk of depression. It takes about 15 minutes to complete. Each item is rated as pass (0) or fail (1). A higher total score indicates worse functioning. KCL has been used as a reliable indicator of daily functioning and progression of disability in Japan National Long-term Care. Taiwan Ministry of Health and Welfare adopted KCL-Taiwan version as an indicator of daily functioning for the use of national-wide disability prevention and delay community-based programs.
General Cognition | up to one month before the start of intervention
  Montreal Cognitive Assessment-Taiwan version (MoCA-T). MoCA-T is in paper-and-pencil format and the maximal score is 30, with higher scores indicating better cognition. MoCA-T total score is adjusted for education effects.
General Cognition | up to one month after the end of intervention
  Montreal Cognitive Assessment-Taiwan version (MoCA-T). MoCA-T is in paper-and-pencil format and the maximal score is 30, with higher scores indicating better cognition. MoCA-T total score is adjusted for education effects.
General Cognition | up to 4 months after the end of intervention
  Montreal Cognitive Assessment-Taiwan version (MoCA-T). MoCA-T is in paper-and-pencil format and the maximal score is 30, with higher scores indicating better cognition. MoCA-T total score is adjusted for education effects.

SECONDARY OUTCOMES:
Functional episodic memory | up to one month before the start of intervention
  Functional episodic memory was assessed by using the event-based task in Miami Prospective Memory Test (MPMT). The participants were asked to pick up an envelope on the desk, get a fixed amount of paper bills from the envelope, give one bill to the examiner and put another one in another envelope when an alarm sounds in 30 minutes later. A total score ranges from 0-9 from three sub-scores of "intention to perform, accuracy, and need for reminders."
Functional episodic memory | up to one month after the end of intervention
  Functional episodic memory was assessed by using the event-based task in Miami Prospective Memory Test (MPMT). The participants were asked to pick up an envelope on the desk, get a fixed amount of paper bills from the envelope, give one bill to the examiner and put another one in another envelope when an alarm sounds in 30 minutes later. A total score ranges from 0-9 from three sub-scores of "intention to perform, accuracy, and need for reminders."
Functional episodic memory | up to 4 months after the end of intervention
  Functional episodic memory was assessed by using the event-based task in Miami Prospective Memory Test (MPMT). The participants were asked to pick up an envelope on the desk, get a fixed amount of paper bills from the envelope, give one bill to the examiner and put another one in another envelope when an alarm sounds in 30 minutes later. A total score ranges from 0-9 from three sub-scores of "intention to perform, accuracy, and need for reminders."
short-term memory and working memory | up to one month before the start of intervention
  Wechsler Adult Intelligence Scale-IV Digit Span subtest (Digits Forward, DF, and Digits Backwards, DB) measure short-term memory (DF) and working memory (DB). Participants listened to a sequence of digits and were asked to recall the sequence correctly (DF) or in reverse-order (DB). Total scores ranged from 2-9 for DF and 2-8 for DB
short-term memory and working memory | up to one month after the end of intervention
  Wechsler Adult Intelligence Scale-IV Digit Span subtest (Digits Forward, DF, and Digits Backwards, DB) measure short-term memory (DF) and working memory (DB). Participants listened to a sequence of digits and were asked to recall the sequence correctly (DF) or in reverse-order (DB). Total scores ranged from 2-9 for DF and 2-8 for DB
short-term memory and working memory | up to 4 months after the end of intervention
  Wechsler Adult Intelligence Scale-IV Digit Span subtest (Digits Forward, DF, and Digits Backwards, DB) measure short-term memory (DF) and working memory (DB). Participants listened to a sequence of digits and were asked to recall the sequence correctly (DF) or in reverse-order (DB). Total scores ranged from 2-9 for DF and 2-8 for DB
Attention and executive Functioning | up to one month before the start of intervention
  Attention and executive Functioning was measured by Color Trail Test Part 1 (CTT-1)(attention) and Part 2 (CTT-2) (executive function) (D'Elia, Satz, Uchiyama, & White, 1996). Participants were asked to connect 25 numbered circles as quickly as possible. Their tests are timed in seconds. The shorter time indicates better performance.
Attention and executive Functioning | up to one month after the end of intervention
  Attention and executive Functioning was measured by Color Trail Test Part 1 (CTT-1)(attention) and Part 2 (CTT-2) (executive function) (D'Elia, Satz, Uchiyama, & White, 1996). Participants were asked to connect 25 numbered circles as quickly as possible. Their tests are timed in seconds. The shorter time indicates better performance.
Attention and executive Functioning | up to 4 months after the end of intervention
  Attention and executive Functioning was measured by Color Trail Test Part 1 (CTT-1)(attention) and Part 2 (CTT-2) (executive function) (D'Elia, Satz, Uchiyama, & White, 1996). Participants were asked to connect 25 numbered circles as quickly as possible. Their tests are timed in seconds. The shorter time indicates better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Ling-Hui Chang, Ph.D, Study Chair — National Cheng Kung University
Locations (1):
- National Cheng-Kung University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mao HF, Tsai AY, Chang LH, Tsai IL. Multi-component cognitive intervention for older adults with mixed cognitive levels: implementation and preliminary effectiveness in real-world settings. BMC Geriatr. 2021 Oct 12;21(1):543. doi: 10.1186/s12877-021-02489-z. PMID 34641803